CLINICAL TRIAL: NCT05900024
Title: An Open-Label, Single-Group Study to Evaluate the Effect of Funk It Cycle Bites on PMS
Brief Title: A Study to Evaluate the Effect of Funk It Cycle Bites on PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Funk It Wellness (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FunkItWellness
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cycle Bites (Experimental): Participants will consume 1 Cycle Bite per day.
  Interventions: Other: Funk It Cycle Bites

INTERVENTIONS:
Other: Funk It Cycle Bites — The intervention product contains: Organic Pumpkin Seed Butter, Prebiotic Agave Inulin, Organic Flax Seed, Organic Oat Flour, Organic Ginger, Quinoa Sprouts, Crispy Red Rice, Organic Cacao Nibs, Sunflower Seed Butter, Organic Reishi Mushroom, Organic Amaranth Seeds, Dates, Organic Button Mushroom, Acai Berry, Amla Fruit, Goji Berry, Pomegranate, Cranberry, Acerola (Cherry Juice), Rosemary Extract, Vitamin E (Mixed Tocopherols), Organic Vanilla Extract, Sea Salt, Cinnamon, Naturally Sourced Potassium Sorbate.

SUMMARY:
This is a virtual, open-label, single-group study that will last 4 menstrual cycles. All participants will complete a questionnaire at the end of their first period after enrolling (baseline/non-intervention cycle 1), then proceed to take the product daily and complete questionnaires at the end of their next 3 periods (intervention cycles 1, 2, and 3). The study will involve 30 female participants with regular menstrual cycles who experience PMS.

Questionnaires will be used to monitor menstrual pain/cramps, energy levels, mood, and hormonal acne experienced before and during the menstrual cycle. Likert scale responses will be statistically compared from baseline to each check-in. Participant responses on product feedback will be presented as % scores.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-40
* Have a regular menstrual cycle (every 21-35 days).
* Suffer from mild to moderate menstrual pain.
* May experience mood swings and/or hormonal acne related to the menstrual cycle.
* Otherwise generally healthy.
* Willing to consume the test product with a ginger flavor.
* Willing to refrain from taking any other supplements or prescription medications that may target the menstrual cycle or premenstrual syndrome (PMS) symptoms throughout the study period.
* Willing and able to adhere to the study protocol, including taking supplements at the required times and completing questionnaires via the technology portal.
* Able to communicate in English.
* Participants must provide written informed consent (ICF).

Exclusion Criteria:

* Any unstable or uncontrolled medical or psychiatric illness.
* Any uncontrolled chronic disease or condition that would prevent full participation in the study protocol.
* A history of polycystic ovary syndrome (PCOS), endometriosis, premenstrual dysphoric disorder (PMDD), or undiagnosed vaginal bleeding.
* Are taking hormonal contraception or exogenous sex hormones (estrogen, testosterone, progesterone), or have taken hormonal contraception or exogenous hormones in the past 6 months.
* Are taking any prescription medication or supplements that target the menstrual cycle or PMS symptoms.
* Are pregnant, breastfeeding, trying to become pregnant, or have been pregnant in the past 12 months.
* Have any known severe allergic reactions, or any allergies of any severity to any of the test product's ingredients.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of premenstrual syndrome. [Time Frame: Baseline to Month 4] | 4 months
  Survey-based assessment of symptoms using the Premenstrual Symptoms Screening Tool (PSST). Responses will be gathered using a 4-point Likert scale.
Changes in acne. [Time Frame: Baseline to Month 4] | 4 months
  Survey-based assessment of acne using the Acne Quality of Life (Acne-QOL) scale. Responses will be gathered using a 5-point Likert scale.
Changes in pain levels, including menstrual cramps. [Time Frame: Baseline to Month 4] | 4 months
  Survey-based assessment of acne using the Numerical Pain Rating Scale, a 0-10 point rating scale.
Changes in mood stability. [Time Frame: Baseline to Month 4] | 4 months
  Survey-based assessment using study-specific questionnaires. Responses will be gathered using a 5-point Likert scale.
Changes in energy levels. [Time Frame: Baseline to Month 4] | 4 months
  Survey-based assessment using study-specific questionnaires. Responses will be gathered using a 5-point Likert scale.

SECONDARY OUTCOMES:
Participant enjoyment of the product. | 4 months
  Survey-based assessment using study-specific questionnaires. Responses will be gathered using a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided